CLINICAL TRIAL: NCT03724474
Title: Integrating Mobile and Wearable Technology to Promote Physical Activity and Sleep Among Midlife Adults: the Bio-Behavioral Systems to Motivate and Reinforce Heart Health (BeSMART) Trial
Brief Title: SMART Technology to Promote Heart Health in Midlife Adults
Acronym: BeSMART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Delaware (Other)
Collaborators: Northern Arizona University (Other)
Responsible Party: Principal Investigator, Greg Dominick, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1168721-1
Record Dates: First submitted 2018-10-04; First posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Physical Activity; Poor Quality Sleep; Hypertension
Keywords: Physical Activity; Sleep; Smartphones; Wearable Activity Monitors; Smart Coaches
MeSH Terms: conditions — Motor Activity; Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized Pretest-Posttest Control Group Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Be SMART Condition (Experimental): Subjects randomly assigned to the Be SMART condition (n=30) will first meet with a credentialed health coach to help create personally relevant weekly, short-term (6-weeks) and long-term (12-weeks) PA and sleep goals, and an initial action and coping plan. At 6- weeks (study mid-point), Be SMART subjects will complete a short telephonic "booster" session with the health coach. Throughout the 12-week intervention, our agent-based feedback system will communicate weekly messages via short message service (SMS) based on their weekly goal achievement, informed by the continuous collection of their Fitbit data. In addition, subjects in the Be SMART condition will also take their morning blood pressure using a blue-tooth enabled device that wirelessly sends this data to the Be SMART server.
  Interventions: Behavioral: Be SMART
- Fitbit Only Condition (Active Comparator): Subjects who are randomly assigned to the active control condition (n=30) will receive a Fitbit device and wireless blood pressure monitor (same as Be SMART condition). However, subjects in the Fitbit Only condition will not meet with a health coach for establishing SMART goals and creating an action/coping plan, nor will Fitbit Only subjects receive any feedback messages or prompts from the Be SMART server, although data from their Fitbit devices will be continuously collected throughout the q12 week intervention.
  Interventions: Behavioral: Be SMART

INTERVENTIONS:
Behavioral: Be SMART — The behavioral intervention will examine 12-week changes in sleep metrics and physical activity, compared to baseline measures, between subjects randomly assigned to a treatment (Be SMART) and an active control (Fitbit Only) condition (n=30, respectively).

SUMMARY:
This study aims to increase weekly minutes of moderate-to-vigorous physical activity and improve sleep quality in a sample of mid-life adults between ages 50 and 64 years.

DETAILED DESCRIPTION:
This 2-year study will develop, test, and refine a cloud-based feedback system, and evaluate the impact of a 3 month randomized controlled feasibility pilot intervention - the Bio-behavioral systems to Motivate and Reinforce Heart Health trial (Be SMART) on changes in moderate-to-vigorous physical activity (MVPA) and sleep among mid-life adults between ages 50 and 64 years.

Aim 1 will examine the acceptability of the Be SMART system. We will conduct a 6-week proof- of-concept study in 10 mid-life adults to specifically examine recruitment plausibility, adherence and attrition rates, satisfaction, and implementation fidelity.

Aim 2 will quantify the impact of the Be SMART intervention (n=30) on changes in MVPA and sleep metrics compared to a Fitbit-only condition (n=30) among mid-life adults (N=60). Hypothesis 2a: At 3 months, participants in the Be SMART condition will show significantly greater weekly minutes of MVPA compared to the Fitbit-only condition, controlling for baseline. Hypothesis 2b: At 3 months, participants in the Be SMART condition will be significantly more likely to report adequate sleep duration, shorter sleep latency, and earlier sleep timing, compared to the Fitbit-only condition, controlling for baseline.

Aim 3 will explore the extent to which changes in MVPA and sleep metrics impact blood pressure changes among mid-life adults (N=60). Secondly, this study will quantify the extent to which Be SMART participants (n=30) achieve their weekly goals and if goal achievement impacts changes in blood pressure at 3 months. Hypothesis 3a: Changes in MVPA and sleep metrics will be related to changes in blood pressure. Hypothesis 3b, the degree of goal achievement will be related to changes in blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* 50-64 years of age
* Prehypertensive (120/80 mmHg - 139/89 mmHg) or stage 1 hypertensive (140/90 mmHg - 159/99 mmHg)
* Physically inactive (<100 minutes of MVPA in the previous week)
* Report insufficient sleep duration (<6 hours/night on >7 nights in the past month)
* Own a smartphone
* Non-smoker
* No signs or symptoms of chronic disease
* Have no chronic pain
* Have no major depressive disorder, general anxiety disorder, or sleep disorder
* Do not work alternating day-night shifts
* Medical clearance obtained from individual's physician

Exclusion Criteria:

* Younger than 50 years; older than 64 years
* Not prehypertensive or blood pressure is >159/99 mmHg
* Physically active (>100 min of MVPA in the previous week)
* Report sufficient sleep duration (>6 hours/night on 7 or more nights in the past month)
* Does not own a smartphone
* Current smoker
* Report signs/symptoms of chronic disease
* Experiences chronic pain
* Have major depressive disorder, general anxiety disorder, or sleep disorder
* Works alternating day and night shifts
* Medical clearance not obtained from individual's physician

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Change in weekly minutes of moderate-to-vigorous physical activity over 12 weeks | 12 weeks
  Participants will wear an accelerometer for 7 consecutive days at baseline and 12 weeks to assess physical activity intensity (e.g. light, moderate, vigorous)